CLINICAL TRIAL: NCT02722278
Title: A Phase 3, Randomized, Active-controlled, Open-label Study of the Safety and Efficacy of Oral Testosterone Undecanoate (TU) in Hypogonadal Men
Brief Title: A Study of Oral Testosterone Undecanoate (TU) in Hypogonadal Men
Acronym: inTUne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CLAR-15012
Record Dates: First submitted 2016-02-15; First posted 2016-03-29 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Testosterone Undecanoate (Experimental): Approximately 135 subjects will receive oral TU treatment during the study for approximately 3.5 months. Subjects randomly assigned to the oral TU treatment group will begin treatment at a dose of 237 mg TU twice daily (BID).
  Interventions: Drug: Oral Testosterone Undecanoate
- Axiron Testosterone Topical Solution (Active Comparator): Subjects randomly assigned to the Axiron treatment group will begin treatment at a dose of 60 mg every morning.
  Interventions: Drug: Axiron Testosterone Topical Solution

INTERVENTIONS:
Drug: Oral Testosterone Undecanoate — Subjects assigned to oral TU treatment will begin at 237 mg TU twice daily. Serial PK samples over 24 hours will be obtained after 21 days and 56 days of treatment. Dose adjustments may be made on Day 35 and Day 70, based on the T Cavg results obtained at Day 21 and Day 56, respectively. Dose will be increased if Cavg < 350 ng/dL, decreased if > 800 ng/dL and maintained if Cavg = 350 ng/dL to 800 ng/dL.
  Other Names: Oral TU
  Arms: Oral Testosterone Undecanoate
Drug: Axiron Testosterone Topical Solution — Subjects assigned to Axiron treatment will begin at 60 mg Axiron every morning. Axiron is applied to the axilla only.
  Serial PK samples over 24 hours will be obtained after 21 days and 56 days of treatment. Dose adjustments may be made on Day 35 and Day 70, based on the T Cavg results obtained at Day 21 and Day 56, respectively. Dose will be increased if Cavg < 350 ng/dL, decreased if > 800 ng/dL and maintained if Cavg = 350 ng/dL to 800 ng/dL.
  Other Names: Axiron solution
  Arms: Axiron Testosterone Topical Solution

SUMMARY:
A Phase 3, Randomized, Active-controlled, Open-label Study of the Safety and Efficacy of Oral Testosterone Undecanoate (TU) in Hypogonadal Men

DETAILED DESCRIPTION:
This is a multicenter, Phase 3, randomized, open-label, active-comparator group, efficacy (based on Cavg of T), and safety study in adult hypogonadal male subjects. Enrollment is based on criteria designed to select the general population of hypogonadal men. Study drug doses will be titrated using a dose-titration algorithm based on total T Cavg. Subjects may be androgen treatment-naïve or washed out of prior androgen replacement therapies.

Subjects must have 2 total T levels < 300 ng/dL based on 2 blood samples obtained in the morning (AM) on 2 separate days approximately 7 days apart.

Approximately 180 subjects will be randomly assigned to receive open-label treatment in a 3:1 ratio of oral TU to Axiron (ie, approximately 135 subjects will be randomly assigned to oral TU and approximately 45 subjects will be randomly assigned to Axiron topical solution). Subjects who complete the study will receive approximately 105 days of treatment. Dose titrations will be based on the T Cavg from serial PK sampling obtained on day 21 and 56 of treatment. Primary efficacy will be based on percentage of subjects within eugonadal range at Visit 7.

A subset of approximately 30 subjects will participate in a cosyntropin stimulation test on Day 1 (before administration of study drug) and Day 106 after the last 24-hour PK sample has been drawn.

ELIGIBILITY:
Inclusion Criteria:

1. Man 18 to 65 years of age, inclusive, with hypogonadism as defined by 2 AM total T values of <300 ng/dL drawn on 2 separate days ([approximately 7 days apart]).
2. Adequate venous access
3. Must be naïve to androgen-replacement therapy or washed out of prior androgen replacement therapies; willing to cease current T treatment or currently not be taking T treatment. Subjects must remain off all forms of T, except for dispensed study drug, throughout the entire study.
4. Subjects on replacement therapy for hypopituitarism or multiple endocrine deficiencies must be on stable doses of thyroid hormone and adrenal replacement hormones for at least 14 days before Screen 1.
5. Voluntarily given written informed consent to participate in this study.

Exclusion Criteria:

1. Received oral topical, intranasal, or buccal T therapy within the previous 2 weeks, intramuscular T injection of short-acting duration within the previous 4 weeks, intramuscular T injection of long-acting duration within the previous 20 weeks, or T implantable pellets within the previous 6 months.
2. Received oral TU in a previous Clarus-sponsored investigational study.
3. Significant intercurrent disease of any type; in particular, liver, kidney, uncontrolled or poorly controlled heart disease, including hypertension, congestive heart failure or coronary heart disease, or psychiatric-illness, including severe depression.
4. Recent (within 2 years) history of stroke, transient ischemic attack, or acute coronary event.
5. A mean of the triplicate assessment of systolic blood pressure (sBP) > 150 mm Hg and/or diastolic blood pressure (dBP) > 90 mm Hg at screening.
6. Recent (within 2 years) history of angina or stent (coronary or carotid) placement.
7. Untreated, severe obstructive sleep apnea.
8. Clinically significant abnormal laboratory values (serum transaminases > 2 × ULN, serum bilirubin > 1.5 × ULN and serum creatinine > 1.5 × ULN).
9. Hematocrit (HCT) value of < 35% or > 48%.
10. Has a history of polycythemia, either idiopathic or associated with testosterone replacement therapy (TRT).
11. Glycosylated hemoglobin (A1C) > 8.5%.
12. BMI ≥ 38 kg/m2.
13. If receiving the following medications:

    * Has been on stable doses of lipid-lowering medication for < 3 months;
    * Has been on stable doses of oral medication for diabetes for < 2 months; or
    * Has been on stable doses of antihypertensive medication for < 3 months.
14. Abnormal prostate digital rectal examination (palpable nodules), elevated Prostate Specific Antigen (serum PSA > 4.0 ng/mL), International Prostate Symptom Score (I-PSS) > 19 points at screening, and/or history of, or current or suspected, prostate cancer.
15. History of, or current or suspected, breast cancer.
16. History of abnormal bleeding tendencies or thrombophlebitis unrelated to venipuncture or intravenous cannulation within the previous 2 years.
17. Use of dietary supplements such as saw palmetto or phytoestrogens and any dietary supplements that may increase total T, such as androstenedione or dehydroepiandrosterone within the previous 4 weeks.
18. Known malabsorption syndrome and/or current treatment with oral lipase inhibitors and bile acid-binding resins.
19. Inability to refrain from smoking during the confinement periods as required by the individual study center.
20. History of alcohol abuse or any drug substance within the previous 2 years.
21. Poor compliance or unlikely to keep clinic appointments.
22. Has received any drug as part of another research study within 30 days of initial dose administration in this study.
23. Donated blood (≥ 500 mL) within the 12-week period before the initial study dose.
24. Currently uses antiandrogens, 5-alpha-reductase inhibitors, estrogens, potent oral CYP3A4 inducers, potent CYP3A4 inhibitors, or long acting opioid analgesics.
25. Unwilling or unable to follow the dietary guidelines for this study, related to taking oral TU with meals that contain approximately 20 to 40 g of fat

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Swerdloff, MD, Principal Investigator — Primary Principal Investigator
Locations (1):
- Multiple Sites in the United States, Northbrook, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data will be shared with all principal investigators following the completion of data analyses

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Testosterone Undecanoate: 166 subjects received oral TU treatment during the study for approximately 3.5 months. Subjects randomly assigned to the oral TU treatment group will begin treatment at a dose of 237 mg TU twice daily (BID).
  Oral Testosterone Undecanoate: Subjects assigned to oral TU treatment will begin at 237 mg TU twice daily. Serial PK samples over 24 hours will be obtained after 21 days and 56 days of treatment. Dose adjustments may be made on Day 35 and Day 70, based on the T Cavg results obtained at Day 21 and Day 56, respectively. Dose will be increased if Cavg < 350 ng/dL, decreased if > 800 ng/dL and maintained if Cavg = 350 ng/dL to 800 ng/dL.
- Axiron Testosterone Topical Solution: 56 subjects were randomly assigned to the Axiron treatment group and began treatment at a dose of 60 mg every morning.
  Axiron Testosterone Topical Solution: Subjects assigned to Axiron treatment will begin at 60 mg Axiron every morning. Axiron is applied to the axilla only.
  Serial PK samples over 24 hours will be obtained after 21 days and 56 days of treatment. Dose adjustments may be made on Day 35 and Day 70, based on the T Cavg results obtained at Day 21 and Day 56, respectively. Dose will be increased if Cavg < 350 ng/dL, decreased if > 800 ng/dL and maintained if Cavg = 350 ng/dL to 800 ng/dL.
Period: Overall Study
Arm/Group | Oral Testosterone Undecanoate | Axiron Testosterone Topical Solution
Started | 166 | 56
Completed | 154 | 49
Not Completed | 12 | 7
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — High PSA pre-study/ not eligible | 0 | 1
Not completed — Subject declined after tx assignment | 0 | 1
Not completed — Site closure not study related | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Axiron Testosterone Topical Solution: Subjects randomly assigned to the Axiron treatment group will begin treatment at a dose of 60 mg every morning.
  Axiron Testosterone Topical Solution: Subjects assigned to Axiron treatment will begin at 60 mg Axiron every morning. Axiron is applied to the axilla only.
  Serial PK samples over 24 hours will be obtained after 21 days and 56 days of treatment. Dose adjustments may be made on Day 35 and Day 70, based on the T Cavg results obtained at Day 21 and Day 56, respectively. Dose will be increased if Cavg < 350 ng/dL, decreased if > 800 ng/dL and maintained if Cavg = 350 ng/dL to 800 ng/dL.
- Total: Total of all reporting groups
Arm/Group | Oral Testosterone Undecanoate | Axiron Testosterone Topical Solution | Total
Number analyzed (Participants) | 166 | 56 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 160 | 54 | 214
  >=65 years | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (9.08) | 53.4 (7.86) | 52 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 166 | 56 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 15 | 40
  Not Hispanic or Latino | 141 | 41 | 182
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 11 | 40
  White | 133 | 42 | 175
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 166 | 56 | 222

OUTCOME MEASURES:

1. Primary Outcome: Number of Oral TU Treated Subjects Who Have a Total T Cavg in the Eugonadal Range of 252 to 907 ng/dL at Visit 7
Time Frame: Day 105
Population: Intent-to-treat study population All subjects randomized to either Oral TU or Axiron
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Testosterone Undecanoate | Axiron Testosterone Topical Solution
Number analyzed (Participants) | 166 | 56
Participants | 145 | 48

2. Other Pre Specified Outcome: Number of Participants With Post-stimulation Cortisol Level of >18 ug/dL at Visit 8
Description: Compare the Oral TU-treated subjects and the Topical Axiron®-treated subjects with respect to number of subjects in the cosyntropin stimulation test substudy with a normal maximum post-stimulation (cosyntropin stimulation) cortisol level at Visit 8.
Time Frame: Approximately 4.5 months
Measure: Count of Participants; unit: Participants
Groups:
- Oral TU Cosyntropin Substudy Subjects: Subjects receiving Oral TU participating in cosyntropin substudy
Arm/Group | Oral TU Cosyntropin Substudy Subjects | Axiron Cosyntropin Substudy Subjects
Number analyzed (Participants) | 24 | 8
Participants | 19 | 8

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Oral Testosterone Undecanoate | Axiron Testosterone Topical Solution
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/166 | 0/55
Other Adverse Events (participants affected / at risk) | 31/166 | 8/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Testosterone Undecanoate (N=166) | Axiron Testosterone Topical Solution (N=55)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periumbilical abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Testosterone Undecanoate (N=166) | Axiron Testosterone Topical Solution (N=55)
High Density Lipoprotein Decreased (Investigations) | 5 (5) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 1 (1)
Prostatic specific antigen increased (Investigations) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 0 (0)
Atypical pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Haematocrit Increased (Investigations) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Hypertension (Vascular disorders) | 5 (5) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 3 (3) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Nerve Compression (Nervous system disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Pelvic Facture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Libido increases (Psychiatric disorders) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Application site pain (General disorders) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1)
Infusion site thrombosis (General disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days